CLINICAL TRIAL: NCT03883256
Title: Effects of High Flow Nasal Cannula on Exercise Endurance in Patients With COPD
Brief Title: High Flow Nasal Cannula on Exercise Endurance in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chen Yen-Huey, assistant professor, Chang Gung University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 201800540A3
Record Dates: First submitted 2019-03-10; First posted 2019-03-20 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: COPD
Keywords: High flow nasal cannula oxygen; exercise performance; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal cannula (Active Comparator): Subjects perform a constant-load exercise test with high flow nasal cannula oxygen device.
  Interventions: Device: high flow nasal cannula
- nasal cannula (Active Comparator): Subjects perform a constant-load exercise test with nasal cannula oxygen device.
  Interventions: Device: nasal cannula

INTERVENTIONS:
Device: high flow nasal cannula — High flow nasal cannula is a device that delivered heated and humidified high flow gases to at or near body temperature to avoid drying and possible injury to the nasal mucosa. In this study, subjects perform a constant-load exercise test with high flow nasal cannula.
  Arms: high flow nasal cannula
Device: nasal cannula — Nasal cannula is a device that delivered oxygen to patients. In this study, subjects perform a constant-load exercise test with nasal cannula.
  Arms: nasal cannula

SUMMARY:
Ventilation limitation has a significant adverse effects on cardiovascular function and cerebral oxygenation during exercise in patients with COPD. High flow nasal cannula (HFNC) has been shown to improve ventilation by washing out the anatomical dead space and permitting a better gas exchanges. Moreover, it is able to ensure the desired inspired oxygen fraction (FiO2) even at high level of patient's minute ventilation by minimizing the room air entrainment. The effects of HFNC on exercise performance in terms of hemodynamic changes and exercise endurance in COPD patients remain unclear. The primary purpose of this study is to examine the effects of HFNC on the exercise endurance in COPD patients. The investigator's secondary purpose is to investigate whether HFNC could improve efficiency of ventilation, leading to an improvement of hemodynamic and cerebral oxygenation response.

DETAILED DESCRIPTION:
This is a randomized crossover study. Patients who have been diagnosed as COPD will be recruited from outpatient department. After signing informed consent form, patients undertake an incremental exercise test and two constant load exercise at the 70% of maximum workload achieved at a previous incremental exercise test on arm ergometer in two separate days. The constant load tests will be performed with HFNC and with nasal cannula at the same inhaled oxygen fraction in random order. The hemodynamics CO, SV, EF of all subjects during exercises will be measured by a bioelectrical impedance device (Physioflow), and cerebral oxygenation status (oxygenated hemoglobin (O2Hb), deoxygenated hemoglobin (HHb), total hemoglobin (tHb) was measured by a near infrared spectrophotometer (NIRS).

ELIGIBILITY:
Inclusion Criteria:

1. with diagnosis of COPD
2. OPD patients
3. has no AE (within 1 month)
4. not receiving any O2 therapy at home
5. no smoking or quick

Exclusion Criteria:

1. fever
2. unstable hemodynamics at resting
3. orthopadeic or neurologic problems that limited exercise

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
exercise time with high flow nasal cannula | end of the exercise test in the session of constant-load exercise test with high flow nasal cannula oxygen device
  the total duration that subjects performed constant-load exercise test with high flow nasal cannula oxygen device
exercise time with nasal cannula | end of the exercise test in the session of constant-load exercise test with nasal cannula oxygen device
  the total duration that subjects performed constant-load exercise test with nasal cannula oxygen device

SECONDARY OUTCOMES:
Difference in cardiac output | Baseline and 48 hours after baseline ]
  Difference in end-exercise cardiac output in constant-load exercise test between HFNCO and NC
Difference in stroke volume | Baseline and 48 hours after baseline ]
  Difference in end-exercise stroke volume in constant-load exercise test between HFNCO and NC
Difference in muscle tissue oxygenation | Baseline and 48 hours after baseline ]
  Difference in end-exercise muscle tissue oxygenation in constant-load exercise test between HFNCO and NC
Difference in cerebral tissue oxygenation | Baseline and 48 hours after baseline ]
  Difference in end-exercise cerebral tissue oxygenation in constant-load exercise test between HFNCO and NC

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huey Chen, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taiwan